CLINICAL TRIAL: NCT01571999
Title: A Single-blind, Non-randomized Pharmacokinetic and Safety Study of Single Dose of GSK573719 and GSK573719 + GW642444 Combination in Healthy Subjects and in Subjects With Severe Renal Impairment
Brief Title: Study to Assess the Safety and PK of GSK573719 and GSK573719/GW642444(VI) Combination in Healthy Subjects and Subjects With Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 114636
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: pharmacokinetics; GW642444; GSK573719; vilanterol; renal impairment; safety; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Renal Insufficiency | interventions — vilanterol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Severe renally impaired subjects (Experimental): Approximately 9 subjects will complete each treatment arm
  Interventions: Drug: Inhaled GSK573719; Drug: Inhaled GSK573719/vilanterol
- Matched healthy volunteers (Experimental): Matched to the severe renal impairment subjects based on gender, ethnicity, body mass index (±15%) and age (±5 years). Approximately 9 subjects will complete each treatment arm
  Interventions: Drug: Inhaled GSK573719; Drug: Inhaled GSK573719/vilanterol

INTERVENTIONS:
Drug: Inhaled GSK573719 — All subjects will receive a single dose of GSK573719 (125mcg) in treatment period 1
Drug: Inhaled GSK573719/vilanterol — All subjects will receive a single dose of GSK573719 (125mcg)/vilanterol (25mcg) in treatment period 2

SUMMARY:
This study will assess the safety and pharmacokinetics of inhaled GSK573719 and GSK573719/vilanterol combination in healthy subjects and in subjects with severe renal impairment. The results of the study will provide guidance on the use of this product in subjects with severe renal impairment.

DETAILED DESCRIPTION:
GSK573719 monotherapy and GSK573719/vilanterol combination are currently under development for the treatment of COPD. This study will assess the pharmacokinetics and safety of inhaled GSK573719 and GSK573719/vilanterol (VI) in healthy subjects and in subjects with severe renal impairment. Nine subjects with severe renal impairment (as defined by a Clcr<30mL/min) will be recruited along with healthy control subjects (as defined by a Clcr>80mL/min matched to the severe renal impairment subjects based on gender, ethnicity, body mass index (±15%) and age (±5 years)). The results from this study will provide guidance on the use of GSK573719 and GSK573719/VI in severe renally impaired patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 70 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea or, child-bearing potential and is abstinent or agrees to use one of the contraception methods listed in the protocol for an appropriate period of time prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until follow-up.

* Body weight greater than or equal to 45 kg and body mass index (BMI) within the range 18 - 33 kg/m2 (inclusive)
* Single QTcF less than 450 msec; or QTc less than 480 msec in subjects with Bundle Branch Block.

Healthy Subjects:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin less than or equal to 1.5x Upper Limit of Normal (ULN)
* Creatinine clearance greater than 80mL/min calculated by the Cockcroft-Gault equation using serum creatinine

Renally Impaired subjects:

* ALT less than 2xULN; alkaline phosphatase and bilirubin less than or equal to 1.5xULN
* Creatinine clearance less than 30mL/min calculated by the Cockcroft-Gault equation using serum creatinine.
* Subjects with renal insufficiency must have stable renal function defined as less than or equal to a 25% difference in creatinine clearance assessed on two occasions. Renal function will be based on estimated creatinine clearance (CLcr) calculated by the Cockcroft-Gault equation using serum creatinine obtained on two occasions separated by at least 4 weeks within the last 3 months

Exclusion Criteria:

* Suffered a lower respiratory tract infection in the 4 weeks before the screening visit
* A supine mean heart rate outside the range 40-90 beats per minute (BPM) at screening
* A positive pre-study drug/alcohol screen
* A positive test for HIV antibody
* Current or chronic history of liver disease, including documented cirrhosis or a history consistent with a diagnosis of cirrhosis, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Use of nephrotoxic medications 4 weeks before dosing
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated
* Subjects with smoking history of greater than 10 cigarettes per day or regular use of tobacco- or nicotine-containing products, within 6 months prior to screening
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Healthy Subjects:

* Subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism or excretion of drugs or any previous gastrointestinal (GI) surgery which the investigator considers sufficiently significant to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Urinary tract or bladder infection within 4 weeks of the first scheduled administration of study drug.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units for males or greater than 14 units for females.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.

Renally Impaired Subjects:

* Life expectancy less than 3 months
* Hemoglobin less than 8.5 g/dL (for sites in Hungary), or hemoglobin less than 11.0g/dL (for sites in the Czech Republic)
* Subjects on hemodialysis treatment
* Subjects who, within the past six months, have had a history of significant drug abuse or alcohol abuse
* Subjects who need to take any concomitant medication, either prescribed or overthe- counter, which may in the opinion of the Investigator, interfere in any way with the study procedure or be a safety concern. In particular subjects taking medications that significantly inhibit P450 CYP3A4 (e.g. ketaconazole) must not be included in this study
* If in the opinion of an examining physician an unstable cardiovascular, pulmonary or hepatic condition is present, or any other medical condition which the investigator considers sufficiently serious to interfere with the conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-03-29 (Actual); Primary Completion 2012-06-22 (Actual); Study Completion 2012-06-22 (Actual)

PRIMARY OUTCOMES:
GSK573719 and vilanterol plasma pharmacokinetic parameters | Treatment Period 1 and 2: pre-dose, 5 mins, 15 mins, 30 mins, 1hr, 2hrs, 4hrs, 8hrs, 12hrs, 16hrs, 24hrs
  Including AUC(0-t), AUC(0-t'), Cmax, tmax, AUC(0-24), AUC(0-infinity), tlast, t1/2

SECONDARY OUTCOMES:
GSK573719 urine pharmacokinetic parameters | Treatment Period 1 and 2: 0-4hrs, 4-8hrs, 8-12hrs, 12-24hrs
Vital Signs Measurements | Screening (up to 21 days before dosing), Treatment Period 1 and 2: pre-dose, 5 mins, 15 mins, 30 mins, 1hr, 4hrs, 12hrs, 24hrs, Follow-up (7 to 14 days after last dose)
  Including systolic and diastolic blood pressure and heart rate
Adverse Events | From administration of first dose until follow-up (7 to 14 days after last dose)
Clinical Laboratory Tests | Screening (up to 21 days before dosing), Treatment Period 1 and 2: pre-dose, 24hrs, Follow-up (7 to 14 days after last dose)
  Including clinical chemistry, haematology and urinalysis tests
12-lead ECG measurements | Screening (up to 21 days before dosing), Treatment Period 1 and 2: pre-dose, 5 mins, 15 mins, 30 mins, 1hr, 4hrs, 12hrs, 24hrs, Follow-up (7 to 14 days after last dose)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Prague, Czechia
- GSK Investigational Site, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Mehta R, Hardes K, Brealey N, Tombs L, Preece A, Kelleher D. Effect of severe renal impairment on umeclidinium and umeclidinium/vilanterol pharmacokinetics and safety: a single-blind, nonrandomized study. Int J Chron Obstruct Pulmon Dis. 2014 Dec 18;10:15-23. doi: 10.2147/COPD.S68094. eCollection 2015. PMID 25565796
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114636 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114636?search=study&search_terms=114636#rs
- Available data/document: Study Protocol: 114636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114636 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register